CLINICAL TRIAL: NCT05395065
Title: Evaluation of the Response of Caries Lesions in Dentin After Application of Silver Diamine Fluoride Gel: A Case Series
Brief Title: Silver Diamine Fluoride Gel: Case Series
Acronym: KiruPoderoso
Status: Completed | Type: Observational
Sponsor: Advantage Silver Dental Arrest, LLC (Industry)
Collaborators: Universidad Nacional Del Altiplano Puno (Unknown); University of Washington (Other)
Responsible Party: Sponsor
Other Study IDs: Gel 2022-1
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Dental Caries in Children
Keywords: Silver Diamine Fluoride; Sodium Fluoride Varnish; Dental Caries; Primary Dentition; Peru
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- SDF/FV: Topical Application of 38% silver diamine fluoride and 2.5% sodium fluoride varnish at baseline and 6 months
  Interventions: Device: Silver Diamine Fluoride/Sodium Fluoride Varnish

INTERVENTIONS:
Device: Silver Diamine Fluoride/Sodium Fluoride Varnish — Application of dental caries arresting topical medication
  Other Names: Advantage Silver Dental Arrest 38% Gel; Fluorimax 2.5% Sodium Fluoride Varnish

SUMMARY:
A clinical case series to determine the clinical response of dental caries lesions in primary teeth where 38% silver diamine fluoride gel is applied and cover with 2.5% sodium fluoride varnish. Additionally, to assess parent satisfaction with treatment with 38% silver diamine fluoride.

DETAILED DESCRIPTION:
A clinical case series of 235 children ages 3 and 4 with severe early childhood caries where the lesions are treated with 38% silver diamine fluoride and covered with 2.5% sodium fluoride varnish at baseline and 6 months. The primary objective is to determine the response of dental caries lesions (caries arrest) into the dentin in primary teeth at one year of follow-up. The secondary objective is to assess parent satisfaction with treatment with 38% silver diamine fluoride and 2.5% sodium fluoride varnish.

ELIGIBILITY:
Inclusion Criteria:

* At least one active caries lesion Good general health by parent report

Exclusion Criteria:

* Unable to cooperate with exam or procedure

Ages: 3 Years to 4 Years | Sex: All
Age Groups: Child
Study Population: The children will be recruited from five schools (Centro Educativo Inicial) in Puno, Peru
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Lesion Activity | 5 months
  Caries Lesion Arrest
Lesion Activity | 12 months
  Caries Lesion Arrest

SECONDARY OUTCOMES:
Caries Increment | 5 months
  Caries Increment (d2-4mfs)
Caries Increment | 12 months
  Caries Increment (d2-4mfs)
New Caries Lesions | 5 months
  Rate of New Caries Lesions ((d2-4mfs)
New Caries Lesions | 12 months
  Rate of New Caries Lesions ((d2-4mfs)
Satisfaction with Color Changes in Teeth | 5 months
  Bothered by Color Changes in the teeth (1-10 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Taina Padilla Caceres, DDS, Principal Investigator — Universidad Nacional del Altiplano
Locations (5):
- Peru (5):
  - UGEL Manazo, Puno
  - UGEL Puno 210001 Las Torres, Puno
  - UGEL Puno Magisterial, Puno
  - UGEL San Jose, Puno
  - UGEL Villa del Lago, Puno

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chu CH, Lo EC, Lin HC. Effectiveness of silver diamine fluoride and sodium fluoride varnish in arresting dentin caries in Chinese pre-school children. J Dent Res. 2002 Nov;81(11):767-70. doi: 10.1177/0810767. PMID 12407092
- [Background] Kiesow A, Menzel M, Lippert F, Tanzer JM, Milgrom P. Dentin tubule occlusion by a 38% silver diamine fluoride gel: an in vitro investigation. BDJ Open. 2022 Jan 13;8(1):1. doi: 10.1038/s41405-022-00095-8. PMID 35027545
- [Derived] Padilla Caceres TC, Cervantes-Alagon S, Castillo JL, Vera Reyes CM, Rothen M, Mancl LA, Milgrom P. Using sequential applications of a novel silver diamine fluoride gel and sodium fluoride varnish to arrest severe early childhood caries lesions: A clinical trial with single group assignment. J Am Dent Assoc. 2024 Jun;155(6):526-535. doi: 10.1016/j.adaj.2024.02.013. Epub 2024 Apr 25. PMID 38678451